CLINICAL TRIAL: NCT02103608
Title: Clinical Evaluation of Silk'n Glide for Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Home Skinovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO105306A
Record Dates: First submitted 2014-03-23; First posted 2014-04-04 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2016-09

CONDITIONS: Hirsutism
Keywords: at Home Photo depilation device, Silk'n.
MeSH Terms: conditions — Hirsutism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Percentage of hair reduction (Experimental): This is an open label, prospective study to evaluate safety and efficiency of Silk'n Glide on the face. During the study, the subjects will perform up to 6 face treatments, two weeks apart. The treatment's safety and efficiency will be evaluated at 4 weeks of after last treatment and at 12 weeks after last treatment .
  Interventions: Device: Glide

INTERVENTIONS:
Device: Glide — 6 facial hair reduction treatments with the Glide device, two weeks apart.

SUMMARY:
This is a clinical study to determine the efficacy and safety of the Glide, hair removal photo-depilation device, for removing facial hairs. During the first stage, the subjects will perform up to 6 face treatments, two weeks apart. The treatment's safety and efficiency will be evaluated at 4 weeks of after last treatment and at 12 weeks after last treatment.

DETAILED DESCRIPTION:
Study efficacy assessment:

Comparison of hair counts before treatments to 4 and 12 weeks follow up visits.

Study safety assessment:

1. Reported errors and near errors using the device
2. Device malfunctions which relate to device safety
3. Device related adverse events
4. Non device related adverse events (secondary endpoint)

ELIGIBILITY:
Inclusion Criteria:

1. Presence of unwanted hairs on the face
2. Skin Type I to IV (Fitzpatrick)
3. Adults older than 21 years of age but not more than 60 years of age.
4. Must be either post-menopausal or surgically steri-lized, or using a medically acceptable form of birth control (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or absti-nence).
5. Informed consent agreement by the subject.
6. Willingness to follow the treatment schedule and post treatment care.

Exclusion Criteria:

1. Malignant or pre-malignant pigmented lesions in the area to be treated.
2. Scarring or infection of the area to be treated.
3. Known photosensitivity.
4. Pregnancy or lactating
5. Subjects with Diabetes (Type I or II).
6. Presence of a suntan in the area to be treated.
7. Use of medication known to induce photosensitivity.
8. Subject is on anticoagulative medication or throm-boembolic condition.
9. Subjects with a pacemaker or internal defibrillator.
10. Use of NSAIDS two weeks prior to, and two weeks following the treatment.
11. Subjects that use waxing or other methods of photo-epilation 3 months prior to treatment.
12. Subjects that have been exposed to strong sunlight or an artificial tanning machine during the past 4 weeks
13. Subjects wearing a tattoo or permanent makeup on the area to be treated
14. Subjects with dark brown or black spots, such as large freckles, birth marks, moles or warts on the area to be treated
15. Subjects with Eczema, psoriasis, lesions, open wounds or active infections, such as cold sores in the area to be treated
16. Subjects with history of keloidal scar formation
17. Subjects with history of herpes outbreaks in the area of treatment, unless you have consulted your physician and received preventative treatment before using GlideTM
18. Subjects with epilepsy
19. Subjects using incontinence device, insulin pump, other active devices [NB: Protocol excludes pace-makers and internal defibrillators.]
20. Subjects with a history of skin cancer or areas of po-tential skin malignancies
21. Subjects who have received radiation therapy or chemotherapy treatments within the past 3 months

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Gold, MD, Principal Investigator — Tennessee Clinical Research Center

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Glide Device: Percentage of hair reduction by the Glide device, the subjects will perform up to 6 face treatments, two weeks apart.
Period: Overall Study
Arm/Group | Glide Device
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Glide Device
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Hair count at baseline [Mean (Standard Deviation); unit: hair strands/cm^2] | 22.7 (14.6)

OUTCOME MEASURES:

1. Primary Outcome: 1. Comparison of Hair Counts Before Treatments to 4 and 12 Weeks Follow up Visits.
Description: Hair count is going to be preformed and base line and compare with the count at 4 weeks and 12 weeks. % of hair reducation is going to be calculated.
Time Frame: 4 weeks and 12 weeks post treatment
Population: Individuals who could benefit from hair reduction
Measure: Mean (Standard Deviation); unit: percentage of hair reduction
Arm/Group | Glide Device
Number analyzed (Participants) | 15
percentage of hair reduction
  4 weeks follow up | 83.3 (22.5)
  12 weeks follow up | 78.1 (34.2)

ADVERSE EVENTS:
Arm/Group | Glide Device
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No